CLINICAL TRIAL: NCT00861575
Title: CAD Genotype and Phenotype Cardiac Catheterization Laboratory Registry
Brief Title: Cardiogenomics Registry
Acronym: CGR
Status: Completed | Type: Observational
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: PH05005
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 20 mL of blood are collected and aliquots of whole blood, plasma, serum and buffy coat are stored.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a continuous blood banking study that will archive plasma and blood permitting DNA and plasma analysis at a future date. Subjects are recruited at the time of a clinically required procedure and blood samples are collected and banked and used for future research. The main purpose of this study is to investigate the interaction of multiple phenotypes and genotypes and their impact on cardiovascular disease events and measures of atherosclerosis progression.

ELIGIBILITY:
Inclusion Criteria:

* > 17 years of age
* Undergoing a clinical required cardiovascular procedure
* Agree to donation of blood sample
* Provide written informed consent and Authorization for Use/Disclosure of PHI

Exclusion Criteria:

* < 18 years of age
* Refusal to donate a blood sample
* Refusal to provide written informed consent and Authorization for Use/Disclosure of PHI

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing a clinical required cardiovascular procedure
Sampling Method: Non-Probability Sample
Enrollment: 2601 (Actual)
Dates: Start 2006-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To assess the relationship of multiple phenotypes and genotypes with cardiovascular disease | Yearly

SECONDARY OUTCOMES:
To assess the impact of phenotypes and genotypes of specific patient subgroups (gender, ethnic, family history) on cardiovascular disease | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rinehart, MD, Principal Investigator — Piedmont Healthcare
Locations (1):
- Piedmont Hospital, Atlanta, Georgia, United States